CLINICAL TRIAL: NCT03924648
Title: Endothelial Cell Specific Molecule-1 (Endocan) Levels in Women With Premature Ovarian Insufficiency
Brief Title: Endocan Levels in Women With Premature Ovarian Insufficiency
Acronym: Endocan&POI
Status: Completed | Type: Observational
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Premature Ovarian Failure
Keywords: Premature menopause; Premature ovarian insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency; Menopause, Premature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premature ovarian insufficiency: Idiopatic premature ovarian insufficiency (POI), defined as loss of ovarian function and subsequent amenorrhea before the age of 40.
  Interventions: Other: Endocan levels
- Control: The investigators compared patients with POI to a cohort of age matched healthy controls recruited among women who visited the gynecology clinic for routine examination or from hospital workers. All volunteers for the control group had regular menstrual cycles and no concomitant health problems.
  Interventions: Other: Endocan levels

INTERVENTIONS:
Other: Endocan levels — Venous blood sample from the antecubital veins for measuring serum concentration of Endocan. The serum endocan level was measured using a commercially available ELISA kit, which is produced to detect human endocan levels with high sensitivity and specificity (Elabscience Biotechnology Inc., Houston, TX, USA). The endocan measurements were performed in accordance with company's protocol.

SUMMARY:
Objective: To evaluate serum endocan levels in women with premature ovarian insufficiency (POI) and to compare the results with those of healthy subjects.

Methods: This prospective study included 38 women with idiopathic POI and 39 controls. The blood for analysis was obtained at the early follicular phase of the menstrual cycle and serum endocan levels were measured using a commercially available ELISA kit. Follicle-stimulating hormone (FSH), estradiol, and anti-mullerian hormone (AMH) were measured at the same time. The continuous values were evaluated using Student's t-test, and categorical values were evaluated using the Chi-square test. P values < .05 were accepted as significant.

DETAILED DESCRIPTION:
Study design This was an observational prospective cohort study conducted at Obstetrics and Gynecology Department of Cengiz Gokcek Obstetrics and Children's Hospital between July and December 2018. Seventy-seven women were enrolled in the study in two groups. All patients gave their oral and written informed consent before their inclusion in the study. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2018/64). The study strictly adhered to the principles of the Declaration of Helsinki.

Data collection and Study intervention:

At enrollment, for both groups, we collected data about age, height, weight, BMI, age of menarche, obstetrics history, history of smoking, regular exercise and family history of POI. The investigators defined that POI period is a time from diagnosis to admission. At enrolment, all patients underwent vaginal ultrasonography for the assessment of antral follicle count (AFC) and venous blood sample from the antecubital veins for measuring serum concentration of Endocan, Follicle-stimulating hormone (FSH), E2, anti-mullerian hormone (AMH) and complete blood count (CBC). In control subjects venous blood samples and AFC were collected during the early follicular phase of the menstrual cycle (2nd to 5th days) in the morning (between 08.00 and 09.00 h). In the POI group, measurements were repeated with 4-week intervals. AMH was not measured in the control group. AFC were assessed through vaginal ultrasonography by the same author (Mindray DC-7T ultrasound machine, Shenzen-Mindray Bio-Medical Electronics Co. Ltd., China). Blood samples were separated by centrifugation for 10 minutes at 1500 g after clotting for 30 minutes at room temperature. The serum samples were subsequently stored in aliquots at -80°C prior to the analysis of endocan. The serum endocan level was measured using a commercially available enzyme-linked immunosorbent assay (ELISA) kit, which is produced to detect human endocan levels with high sensitivity and specificity (Elabscience Biotechnology Inc., Houston, TX, USA). The endocan measurements were performed in accordance with company's protocol. The kit uses the sandwich ELISA principle. A biotinylated detection antibody specific for human ESM1 (endocan) and avidin-horseradish peroxidase conjugate were used in the measurement. Spectrophotometry at a wave length of 450 ± 2 nm was used in the detection of optical density, which is proportional to the concentration of human endocan level. The intra- and inter-assay variation coefficients were 6.36% and 6.09%, respectively.

Endpoints of the study:

The primary endpoint in this analysis was to compare endocan levels in POI group and control group. The secondary endpoint was to compare endocan levels in POI group for POI period. Tertiary endpoint was to compare the endocan levels in both groups according to the births.

The normality of distribution of continuous variables was tested using the Shapiro-Wilk test. To compare numerical variables between 2 groups, Student's t-test (for normal data) or the Mann-Whitney U test (for non-normal data) was performed. The Chi-square test was used to assess the relationship between categorical variables, and Spearman's rank correlation coefficients were used to assess the relationship between non-normal numeric data. Frequency, percentage (%) and mean ± standard deviations (mean ± SD) are given as descriptive statistics. Statistical analysis was performed using the SPSS for Windows version 24.0 software package, and p valued < 0.05 were accepted as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic POI
* age-matched healthy controls.

Exclusion Criteria:

* Women with evidence for karyotypic, metabolic, toxic, or iatrogenic cause of the ovarian insufficiency
* Any women who use any medication for POI treatment,
* Women who had fever
* Women who had any Cardiovascular diseases

Ages: 18 Years to 39 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Premature ovarian insufficiency (POI), defined as loss of ovarian function and subsequent amenorrhea before the age of 40
Study Population: The investigators consecutively recruited 38 subjects with idiopathic POI, and 39 healthy patients were selected for the control group. The investigators included patients with the diagnosis of idiopathic POI independently from the year of diagnosis. The investigators compared patients with POI to a cohort of age matched healthy controls recruited among women who visited the gynecology clinic for routine examination or from hospital workers. All participants for the control group had regular menstrual cycles and no concomitant health problems.
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this analysis was to compare endocan levels in POI group and control group. | 1 day
  The primary endpoint in this analysis was to compare endocan levels in POI group and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ovayolu, MD, Principal Investigator — Cengiz Gokcek WCH
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maclaran K, Panay N. Current concepts in premature ovarian insufficiency. Womens Health (Lond). 2015 Mar;11(2):169-82. doi: 10.2217/whe.14.82. PMID 25776291
- [Background] de Kat AC, Verschuren WM, Eijkemans MJ, Broekmans FJ, van der Schouw YT. Anti-Mullerian Hormone Trajectories Are Associated With Cardiovascular Disease in Women: Results From the Doetinchem Cohort Study. Circulation. 2017 Feb 7;135(6):556-565. doi: 10.1161/CIRCULATIONAHA.116.025968. PMID 28153992

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-28): https://cdn.clinicaltrials.gov/large-docs/48/NCT03924648/Prot_SAP_000.pdf